CLINICAL TRIAL: NCT02032238
Title: Clinical Efficacy of Bevacizumab Combined With Navigated Laser in Patients With Clinically Significant Macula Edema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of anticipated participants was not achieved
Sponsor: OD-OS GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAVNAV-2
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Clinically Significant Macular Edema

STUDY DESIGN:
Masking Description: no masking

ARMS (2):
- laser photocoagulation with bevacizumab (Experimental): Combining laser photocoagulation and Anti-VEGF Injections in a pre-defined manner
  Interventions: Device: laser photocoagulation
- Bevacizumab, no laser photocoagulation (No Intervention): patients receive Anti-VEGF injections (Bevacizumab) only

INTERVENTIONS:
Device: laser photocoagulation — Standard bevacizumab Injections will be combined with laser photocoagulation in a pre-defined manner
  Arms: laser photocoagulation with bevacizumab

SUMMARY:
Asses efficacy of navigated laser in reducing the number of anti-VEGF injections as a prospective study using Bevacizumab.

DETAILED DESCRIPTION:
The purpose of this is study is to assess the efficacy of navigated laser treatment in reducing the number of anti-VEGF injections required to maintain visual gain obtained after Bevacizumab compared to Bevacizumab alone in patients with clinically significant macular edema (CSME).

This will be prospective, active-controlled study using Bevacizumab (Genentech, South San Francisco CA) for intravitreal injections. Retinal photocoagulation will utilize the Navilas Laser System (OD-OS GmbH, Teltow, Germany), which is an approved indication for this device.

ELIGIBILITY:
Inclusion Criteria:

* CSME and Diagnosis of diabetes mellitus
* Able and willing to provide informed consent prior to any study-related procedures
* Central foveal thickness > 250 microns at baseline
* Best corrected visual acuity between 20/400 and 20/40
* Willing and able to comply with clinic visits and study-related procedures
* U.S. patients will be required to have a Health Insurance Portability and Accountability Act (HIPAA) authorization; in other countries, as applicable according to national laws

Exclusion Criteria:

* - Macular edema is considered to be due to a cause other than diabetic macular edema.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., macular ischemia, vitreomacular traction, foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition).
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.)
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of treatment for diabetic macular edema at any time in the past 4 months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, anti-VEGF drugs, or any other treatment).
* History of panretinal (scatter) photocoagulation (PRP) within 4 months prior to enrollment.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization. 13
* History of YAG capsulotomy performed within 2 months prior to randomization.
* Aphakia.
* Intraocular pressure >= 25 mmHg.
* History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: history of angle-closure glaucoma is not an exclusion criterion).
* History of steroid-induced intraocular pressure (IOP) elevation that required IOP-lowering treatment.
* Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control)
* Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry
* Known allergy to any component of the study drug
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
* Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.
* Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
* Systemic anti-vascular growth factor (anti-VEGF) or pro-VEGF treatment within 4 months prior to randomization 14
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months.
* Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the first 12 months of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, Study Director — OD-OS
Locations (1):
- Eye and Ear Infirmary, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser Photocoagulation With Bevacizumab | Bevacizumab, no Laser Photocoagulation
Started | 12 | 0 (Study Terminated due to slow enrollment, no subjects enrolled in this study arm)
Completed | 10 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Combination With Navigated Laser: Combining photocoagulation and Anti-VEGF Injections in a pre-defined manner
  Navigated laser: Standard Anti-VEGF Injections will be combined with Navigated laser in a pre-defined manner
  Anti-VEGF Injections: Monotherapy
- Monotherapy: patients receive Anti-VEGF Monotherapy
  Anti-VEGF Injections: Monotherapy
- Total: Total of all reporting groups
Arm/Group | Combination With Navigated Laser | Monotherapy | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 6 |  | 6
  >=65 years | 6 |  | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes That Received Retreatment
Time Frame: 12 months
Measure: Number; unit: Percentage of eyes that received retreat
Arm/Group | Combination With Navigated Laser | Monotherapy
Number analyzed (Participants) | 10 | 0
Percentage of eyes that received retreat | 55.56 |

ADVERSE EVENTS:
Arm/Group | Laser Photocoagulation With Bevacizumab | Bevacizumab, no Laser Photocoagulation
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less